CLINICAL TRIAL: NCT00732342
Title: Contingency Management Treatment Duration
Acronym: Duration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 08-053-2; P60AA003510 (NIH)
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Abuse
Keywords: Alcohol Abuse; Contingency Management; Treatment Duration
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): Standard Treatment
- 2 (Experimental): Standard Treatment with Contingency Management for 12 weeks with a 0.5 probability of winning prizes for each negative sample submitted
  Interventions: Behavioral: Contingency Management
- 3 (Experimental): Standard Treatment with Contingency Management for 24 weeks with a 0.34 probability of winning prizes for each negative sample submitted
  Interventions: Behavioral: Contingency Management
- 4 (Experimental): Standard Treatment with Contingency Management for 24 weeks with a 0.5 probability of winning prizes for each negative sample submitted
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Prizes given for targeted behavior of abstinence
  Arms: 2; 3; 4

SUMMARY:
310 alcohol abusing or dependent patients beginning intensive outpatient day treatment at community-based clinics will be randomly assigned to one of four conditions: (a) standard treatment as usual (ST) at the clinic without contingency management (CM); (b) standard treatment with contingency management for 12 weeks with a 0.5 probability of winning prizes for each negative sample submitted; (c) standard treatment with contingency management for 24 weeks with a 0.34 probability of winning prizes for each negative sample submitted; or (d) standard treatment with contingency management for 24 weeks with a 0.5 probability of winning prizes for each negative sample submitted. We expect that contingency management will decrease alcohol use to a greater extent than non-contingency management treatment, and that availability of contingency management for 24 weeks may result in longer term benefits than 12 week exposure to contingency management. This study will be the first to evaluate the effects of probability of winning prizes on response to contingency management.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* current DSM-IV diagnosis of alcohol abuse or dependence
* willing to sign informed consent and able to pass an informed consent quiz

Exclusion Criteria:

* serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, bipolar disorder, severe or psychotic major depression, or suicide risk) on the basis of history or medical examination
* current DSM-IV diagnosis of opioid dependence
* in recovery from pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2008-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
longest duration of negative breath samples submitted | active phase and throughout follow-up phase

SECONDARY OUTCOMES:
subjective reports of alcohol use | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health
Locations (5):
- United States (5):
  - Prospect House, Bridgeport, Connecticut
  - Alcohol and Drug Recovery Centers, Inc., Hartford, Connecticut
  - The Hospital of Central Connecticut at New Britain General, New Britain, Connecticut
  - Morris Foundation, Waterbury, Connecticut
  - Carlson Recovery Center, Springfield, Massachusetts